CLINICAL TRIAL: NCT02012569
Title: A Phase II Randomized, Controlled, Single Blind Study to Evaluate the Haemostatic Efficacy and Safety of TT-173 Applied in the Donor Site of Patients Undergoing Skin Graft
Brief Title: Determine the Haemostatic Efficacy of TT-173, Reducing the Bleeding Time in the Donor Site of Skin Grafting
Acronym: EHTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thrombotargets Europe S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THO-IM_01-CT; 2013-002784-25 (EudraCT Number)
Record Dates: First submitted 2013-11-21; First posted 2013-12-16 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2015-11

CONDITIONS: Burns; Traumatic Lesions
Keywords: skin grafting; elective treatment
MeSH Terms: conditions — Burns | interventions — Hemostasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TT.173 (Experimental): It is applied directly to the bleeding of the donor site
  Interventions: Drug: TT-173
- placebo (Placebo Comparator): It is applied directly to the bleeding of the donor site
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TT-173 — Bleeding of the lesion will be evaluated after each product application and will be recorded as bleeding vs. not bleeding. The product will be applied at 4 times for about 1 minute apart each application after skin graft obtention.
  Other Names: topical hemostatic agent
  Arms: TT.173
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the haemostatic efficacy of TT-173, reducing the bleeding time in the donor site of skin grafting.

DETAILED DESCRIPTION:
As the TT-113 has been cleared for use as a topical hemostatic agent, the proposed study will further investigate the safety and efficacy of TT-113 in the donor site of sking grafting

ELIGIBILITY:
Inclusion Criteria:

* Subjects who signed the informed consent.
* Subjects that have to undergo a skin graft.
* Subjects of both sexes older than 18 years.
* Subjects that present a burn or traumatic skin injury affecting less than 30% of corporal surface.
* Subjects with a platelet count not compatible with pathology.
* Subjects who present haemogram results not indicative of any of the situations mentioned in the exclusion criteria.
* Subjects who present biochemical results not indicative of any of the situations mentioned in the exclusion criteria.
* Subjects who present coagulation parameters not indicative of any of the situations mentioned in the exclusion criteria.
* Women of childbearing age who take contraceptive measures and are willing to maintain them until the end of follow up of this study.
* Women of childbearing age who present a negative test pregnancy at the moment of study inclusion

Exclusion Criteria:

* -Subjects with personal or family history of abnormal hemorrhagic episodes.
* Subjects affected of any kind of congenital or acquired coagulopathies.
* Subjects that present a burn or traumatic skin injury affecting more than 31% of corporal surface.
* Subjects affected of any blood, heart or liver disease, chronic renal failure, severe chronic obstructive pulmonary disease, active oncologic process in the past three months, diabetes type I or who has suffered a stroke.
* Subjects who experienced excessive bleeding after surgical procedures, childbirth or tooth extraction.
* Subjects affected by any acute infectious disease.
* Subjects affected of any systemic disease that may worsen the prognosis if any adverse effect occurs (decompensated type 2 diabetes mellitus, uncontrolled hypertension or severe systemic disease).
* Subjects who should take antiplatelet therapies one week before and 48 hours after the surgery (AAS, trifusal, dipiridamol, clopidogrel, abciximab).
* Subjects with known hypersensitivity or allergy to any component of the drug.
* Subjects who consume abuse drugs excluding cannabis and its derivatives.
* Subjects who are unable to follow or understand properly the instructions and requirements of the study.
* Subjects who are not free to give informed consent or who are mentally incapacitated to the discretion of investigators.
* Subjects who participate or have participated in the past three months in another clinical trial with drug treatment.
* Subjects that are the investigators, collaborators, nurses, center employees or any other person directly related to the development of the protocol.
* Subjects who are positive to HIV or HCV serology, or who present active HBV infection.
* Subjects who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Reducing the bleeding time in the donor site of skin grafting | 10 min

SECONDARY OUTCOMES:
Safety and tolertability | 1 month
  Number of Adverse Events
Systemic absorption of the product | 1 month
  Cmax, Tmax, AUC and bioavailability
Immunogenicity | 1 month
  Antibody concentration

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Rojas, Manager, Study Director — Thrombotargets Europe
Locations (1):
- Thrombotargets Europe, Castelldefels, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lopez-Lopez J, Jane-Salas E, Santamaria A, Gonzalez-Navarro B, Arranz-Obispo C, Lopez R, Miquel I, Arias B, Sanchez P, Rincon E, Rodriguez JR, Rojas S, Murat J. TETIS study: evaluation of new topical hemostatic agent TT-173 in tooth extraction. Clin Oral Investig. 2016 Jun;20(5):1055-63. doi: 10.1007/s00784-015-1586-1. Epub 2015 Sep 15. PMID 26374745
- See also: For more information about this study: Clinical Oral Investigations journal — http://link.springer.com/article/10.1007%2Fs00784-015-1586-1